CLINICAL TRIAL: NCT01454752
Title: Intermittent Parasite Clearance (IPC) in Schools: a Randomised Double-blind Placebo-controlled Trial of the Impact of IPC on Malaria, Anaemia and Cognition Amongst School Children in Kedougou, Senegal
Brief Title: Intermittent Parasite Clearance (IPC) in Schools: Impact on Malaria, Anaemia and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Division Controle Medicale Scolaire, Ministry of Education, Senegal (Unknown); Ministry of Health, Senegal (Other Government); Institut National d'Etude et d'Action pour le Developpement de l'Education, Senegal (Unknown); Cheikh Anta Diop University, Senegal (Other); Institut de Recherche pour le Developpement, Senegal (Other); Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: WT-Clarke-Sen2011
Record Dates: First submitted 2011-10-12; First posted 2011-10-19 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Malaria; Anaemia
Keywords: malaria; anaemia; cognition; intermittent preventive treatment; children; schools; insecticide-treated nets
MeSH Terms: conditions — Malaria; Anemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent parasite clearance (Active Comparator): Children sleeping under a long-lasting insecticidal net (LLIN) receive an additional intermittent preventive treatment for clearance of asymptomatic malaria infection given once a year at the end of the malaria transmission season
  Interventions: Drug: Intermittent parasite clearance
- Control (Placebo Comparator): Children sleeping under a long-lasting insecticidal net (LLIN) receive placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Intermittent parasite clearance — Sulphadoxine-pyrimethamine (500/25mg) according to age, given on day 1; Amodiaquine (200mg) according to age, given daily for 3 days
  Arms: Intermittent parasite clearance
Other: Placebo — Placebo tablets, similar in appearance and taste to active treatment, given daily over 3 days
  Arms: Control

SUMMARY:
Although the risk of malaria is greatest in early childhood, significant numbers of schoolchildren remain at risk from malaria infection, clinical illness and death. By the time they reach school, many children have already acquired some clinical immunity and the ability to limit parasite growth, and thus most infections are asymptomatic and will go undetected and untreated. Asymptomatic parasitaemia contributes to anaemia, reducing concentration and learning in the classroom, and interventions aiming to reduce asymptomatic parasite carriage may bring education, as well as health, benefits.

Intermittent parasite clearance (IPC) delivered through schools is a simple intervention, which can be readily integrated into broader school health programmes, and may usefully supplement the community-distribution of insecticide-treated nets (ITNs) in countries with a policy of universal coverage of nets.

This study seeks to establish whether intermittent parasite clearance undertaken once a year at the end of the malaria transmission season can reduce malaria parasite carriage and anaemia amongst school-going children already using insecticide-treated nets, and its consequent impact on school attendance and performance, in order to assess its suitability for inclusion as a standard intervention in school health programmes in areas of seasonal malaria transmission.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in participating elementary schooled
* provision of parental consent

Exclusion Criteria:

* lack of consent
* chronic conditions which limit regular school attendance
* clinical malaria on the day of scheduled treatment (as defined as febrile, with a positive result in a rapid diagnostic test for malaria).

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 860 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of malaria parasitaemia | 8 weeks after treatment (February 2012)
Prevalence of anaemia (Haemoglobin<11 g/dL) | 8 weeks after treatment (February 2012)

SECONDARY OUTCOMES:
Cognitive performance in tests of sustained attention | 8 weeks after treatment (February 2012)

CONTACTS AND LOCATIONS:
Overall Officials: Sian E Clarke, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Institut de Recherche pour le Developpement, Dakar, Senegal